CLINICAL TRIAL: NCT03368417
Title: A Randomised Controlled Trial to Improve Hypertension Outcomes Using Wireless Home Blood Pressure Monitoring With Automatic Outcome-based Feedback and Financial Incentives
Brief Title: WIreless Monitoring and Financial Incentives for Uncontrolled HYpertension (WIFHY) Study
Acronym: WIFHY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to unforeseen delays and funding issues
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: SingHealth Polyclinics (Other)
Responsible Party: Principal Investigator, Marcel Bilger, Assistant Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSRG13MAY009
Record Dates: First submitted 2017-11-28; First posted 2017-12-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Hypertension
Keywords: Hypertension; Wireless Home Blood Pressure Monitoring; Medication Adherence; Medication Titration; Financial Incentives; Ambulatory Blood Pressure Monitoring
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (Active Comparator): Usual care from SingHealth Polyclinics which includes non-wireless HBPM. In addition, participants will receive a medication event monitoring system and will be on ambulatory blood pressure monitoring at baseline and Month 6.
  Interventions: Other: Usual Care
- Wireless HBPM System (Experimental): Usual care from SingHealth Polyclinics with wireless HBPM system. In addition, participants will receive a medication event monitoring system and will be on ambulatory blood pressure monitoring at baseline and Month 6.
  Interventions: Other: Usual Care; Other: Wireless HBPM System
- Wireless HBPM System and Incentives (Experimental): Usual care from SingHealth Polyclinics with wireless HBPM system and BP monitoring incentives. In addition, participants will receive a medication event monitoring system and will be on ambulatory blood pressure monitoring at baseline and Month 6.
  Interventions: Other: Usual Care; Other: Wireless HBPM System; Behavioral: BP Monitoring Incentives

INTERVENTIONS:
Other: Usual Care — Participants will be advised to measure their BP at least 3 times a week and record their results on a form. The participants will be educated on how to interpret their BP according to standard self-monitoring practice guidelines.
  As part of the study, participants without a HBPM will be provided with the Omron HEM 7130. Adherence to hypertensive medicines will be monitored using the medication event monitoring system eCAP™. In addition, the participants will be asked to undertake ambulatory blood pressure monitoring (using the Welch Allyn ABPM 7100 monitor) at Baseline and Month 6 for a duration of 12 hours, during their waking hours.
Other: Wireless HBPM System — BP will be monitored using the iHealth KN-550BT wireless HBPM and transmitted to the study application via the iHealth mobile application.
  The Wireless HBPM System consists of:
  i) Instant BP feedback: Classification of each BP reading with feedback SMS. CRC will call the patient in case of alarming BP readings.
  ii) Weekly HBPM adherence feedback: Participants receive praise, encouraging, or reminder SMSes.
  iii) Continuous assessment: Based on average BP over the last 4 weeks, participants will be categorized and flagged for the CRC to follow clinical protocols. Protocols include asking patients to immediately come to the clinic, checking for alarm symptoms and discussing adherence over the phone, remote titration, and cancelling 1 clinic visit in case of good BP control.
  Arms: Wireless HBPM System; Wireless HBPM System and Incentives
Behavioral: BP Monitoring Incentives — Participants will receive an intervention identical to those in the Wireless HBPM System, with financial incentives for BP monitoring. This arm is further randomly subdivided into the Instant Reward and Health Capital arms in a 1:1 ratio.
  Instant Reward sub-arm:
  * Participants receive SGD 3 for each day they measure their BP, up to three times per week.
  * Participants do not receive financial incentive if they do not measure their BP.
  Health Capital sub-arm:
  * Participants receive an initial health capital of SGD 72
  * Participants' health capital increases by SGD 6 on each week where they measure their BP on at least 3 different days and decreases weekly by 10% per missing BP reading.
  Arms: Wireless HBPM System and Incentives

SUMMARY:
Hypertension is a major risk factor for cardiovascular morbidity and mortality. Despite the risks of hypertension and availability of effective treatment, a substantial number of patients have uncontrolled Blood Pressure (BP). Systematic reviews have shown that Home Blood Pressure Monitoring (HBPM) produces modest improvements in BP control and that HBPM yields greater benefits when combined with other interventions such as remote titration change or adherence-enhancing strategies.

The investigators propose a Wireless HBPM System comprising of a Wireless Home Blood Pressure Monitor and a Study Application that aims to: provide text messaging on BP advice and reminders on BP management based on BP readings; promote adherence to BP monitoring and adherence to medication; flag patients for counselling on medication adherence and remote titration (by doctor) during in-between visits; cut the response time in case of emergency; and skip polyclinic visits for well-managed patients.

An additional arm will include the the addition of modest financial incentives for participants when they monitor their BP. This arm is subdivided into two sub-arms (Instant Reward and Health Capital) where patients are eligible to receive the same incentive amounts but framed differently.

This study is novel in its comprehensive approach to patient disease self-management and remote provision of medical care, potentially reducing the burden on the health system and improving patient health outcomes.

DETAILED DESCRIPTION:
Hypertension is a major risk factor for cardiovascular morbidity and mortality. The ultimate goal of hypertension treatment is to lower blood pressure (BP) and thereby reduce cardiovascular risk. Despite the risks of hypertension and availability of effective treatment, a substantial number of patients have uncontrolled BP. Systematic reviews have shown that Home Blood Pressure Monitoring (HBPM) produces modest improvements in BP control and that HBPM yields greater benefits when combined with other interventions such as remote titration change or adherence-enhancing strategies.

The effectiveness of HBPM is tempered because many patients with access to home BP monitors fail to regularly measure their BP or respond appropriately to high readings. New technology has made tele-monitoring of patient health feasible and has allowed for measurement and transmission of patient BP and other patient information from the home to a health care provider. An additional strategy to further improve the compliance of the patients with their hypertension management plan is to provide them with a clearer short term benefit, rewarding compliance. For example, those who achieve BP within the target range could receive a financial incentive.

The investigators' strategy to improve the effectiveness of HBPM to reduce BP is to use the full potential of wireless and mobile technology to create automatic feedback loops between the patient and the health care provider. The investigators propose a 6-month randomized controlled trial with 224 hypertensive patients with uncontrolled BP from the SingHealth Polyclinics in Bedok and Marine Parade, Singapore. The proposed trial will be a parallel study with one control arm and two intervention arms in ratio of 2:3:3 with the objective of measuring the incremental effectiveness and cost-effectiveness of an intervention with Wireless HBPM System, with and without financial incentives, compared to non-wireless HBPM alone.

Specifically, the investigators have the following primary aims and hypotheses:

A1: Determine whether a Wireless HBPM System with and without financial incentives is effective at reducing systolic blood pressure (SBP) compared to a non-wireless HBPM that relies on patient self-reporting and best practices (Usual Care, UC).

H1a: The average reduction in SBP at 6 months will be greater for the patients in the intervention arms (Wireless HBPM System with and without Incentives) compared to UC patients.

H1b: The average reduction in SBP at 6 months will be greater for the patients in the Wireless HBPM System with incentives arm compared to those in the Wireless HBPM System without incentives arm.

As well as the following secondary aims and hypotheses:

A2: Determine whether a Wireless HBPM System with and without financial incentives is effective at reducing diastolic blood pressure (DBP) compared to a non-wireless HBPM that relies on patient self-reporting and best practices (Usual Care, UC).

H2a: The average reduction in DBP at 6 months will be greater for the patients in the intervention arms (Wireless HBPM System with and without incentives) compared to UC patients.

H2b: The average reduction in DBP at 6 months will be greater for the patients in the Wireless HBPM System with incentives arm compared to those in the Wireless HBPM System without incentives arm.

A3: Quantify the incremental cost-effectiveness of Wireless HBPM System without incentives compared with UC, and of Wireless HBPM System with incentives compared to Wireless HBPM without Incentives.

H3a: The Incremental Cost-Effectiveness Ratio (ICER) of Wireless HBPM System without incentives compared to UC will be favorable relative to international benchmarks for cost-effectiveness analysis.

H3b: The ICER of Wireless HBPM System with incentives compared to Wireless HBPM System without incentives will be favorable relative to other published RCTs with primary aim of reducing SBP.

A4: Determine whether a Wireless HBPM System with and without financial incentives is effective at decreasing patient non-adherence to BP self-monitoring and hypertensive medicines compared to a non-wireless HBPM that relies on patient self-reporting and best practices (Usual Care, UC).

H4a, H4b: The average number of missing BP measurements (H4a) and percentage of medication doses not taken (H4b) during the last month of the study will be smaller for the patients in the intervention arms (Wireless HBPM System with and without incentives) compared to UC patients.

H4c, H4d: The average number of missing BP measurements (H4c) and percentage of medication doses not taken (H4d) during the last month of the study will be smaller for the patients in the Wireless HBPM System with incentives arm compared to those in the Wireless HBPM System without incentives arm.

A5: Determine whether financial incentives framed as health capital is effective at decreasing patient non-adherence to BP self-monitoring compared to financial incentives framed as a reward.

H5: The average number of missing BP measurements over the intervention period will be smaller for the patients in the Health Capital sub-arm compared to those in the Instant Reward sub-arm.

ELIGIBILITY:
Inclusion Criteria:

* Known hypertensive patients on at least one anti-hypertensive medication
* SBP more than or equal to 140 mmHg or DBP more than or equal to 90 mmHg for patients without diabetes, SBP more than or equal to 140 mmHg or DBP more than or equal to 85 mmHg for patients with diabetes, as verified by the average of the last 2 of 3 BP readings taken, on the day of polyclinic visit, at 3 minutes interval using the Omron HEM-7130
* Aged between 21 to 70 years of age;
* Singaporean citizens or Permanent Residents;
* Able to converse in English or Mandarin;
* Has a compatible smartphone (iOS Versions 8.0 and higher or Android Versions 5.0 and higher) with data plan or regular Wi-Fi access
* Ability to perform self-monitoring of BP as assessed by the CRC
* Expecting to be a patient of Bedok or Marine Parade Polyclinics for the duration of the trial

Exclusion Criteria:

* SBP equal or greater than 180mmHg or DBP equal or greater than 110mmHg, as verified by the average of the last 2 of 3 BP readings taken, on the day of polyclinic visit, at 3 minutes interval using the Omron HEM-7130
* pregnancy
* clinically unstable heart failure
* advanced kidney disease, i.e. eGFR < 30 ml/min
* known liver disease
* Atrial Fibrillation
* underwent Double Mastectomy
* any other major debilitating disease or mental illness that precludes validity of informed consent or would result in the patient being unable to take their BP independently.
* started on angiotensin-converting enzyme inhibitors (ACE inhibitors) or angiotensin- receptor blockers (ARB) within the last 3 months
* on Warfarin or anti-coagulants (e.g. NOACs: Novel Oral Anticoagulants)
* known allergy to epoxy resin
* discharged from hospital within the last 3 months for complications related to hypertension
* newly referred to Specialist Outpatient Clinics (SOCs) or on follow-up for complications related to hypertension
* severe or overt macro albuminuria (urine ACR>30mg/mmol or PCR>0.5)
* confirmed glomerulonephritis
* living in a household where another member has been recruited into the trial

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-01-27 (Actual); Study Completion 2019-01-27 (Actual)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure (SBP) | Between baseline and Month 6
  Change in average SBP between baseline and Month 6 as measured by ambulatory blood pressure monitoring using the Welch Allyn ABPM 7100 monitor. At each time point (baseline and Month 6), ABPM frequency will be set at one BP measurement every 30 minutes for a duration of 12 waking hours, and average SBP will be calculated.

SECONDARY OUTCOMES:
Change in Diastolic Blood Pressure (DBP) | Between baseline and Month 6
  Change in average DBP between baseline and Month 6 as measured by ambulatory blood pressure monitoring using the Welch Allyn ABPM 7100 monitor. At each time point (baseline and Month 6), ABPM frequency will be set at one BP measurement every 30 minutes for a duration of 12 waking hours, and average DBP will be calculated.
Mean weekly number of missing BP readings | during Month 6
  Participants are recommended to take their BP at least 3 times each week. This outcome measures the average weekly number of missing BPs over the last month of the intervention (Month 6).
Mean weekly number of missing BP readings | from Month 1 to Month 6
  Participants are recommended to take their BP at least 3 times each week. This outcomes measure the average weekly number of missing BPs over the entire duration of the intervention.
Mean proportion of antihypertensive medication doses not taken | during Month 6
  Medication adherence will be measured using the medication event monitoring system eCAP™. This outcome measures the proportion of scheduled antihypertensive medications that were not taken by the participant during the last month of the intervention (Month 6).

CONTACTS AND LOCATIONS:
Overall Officials: Dr Marcel Bilger, Principal Investigator — Duke-NUS Graduate Medical School
Locations (2):
- Singapore (2):
  - Marine Parade Polyclinic, Singapore
  - Bedok Polyclinic, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] MacMahon S, Peto R, Cutler J, Collins R, Sorlie P, Neaton J, Abbott R, Godwin J, Dyer A, Stamler J. Blood pressure, stroke, and coronary heart disease. Part 1, Prolonged differences in blood pressure: prospective observational studies corrected for the regression dilution bias. Lancet. 1990 Mar 31;335(8692):765-74. doi: 10.1016/0140-6736(90)90878-9. PMID 1969518
- [Background] Collins R, Peto R, MacMahon S, Hebert P, Fiebach NH, Eberlein KA, Godwin J, Qizilbash N, Taylor JO, Hennekens CH. Blood pressure, stroke, and coronary heart disease. Part 2, Short-term reductions in blood pressure: overview of randomised drug trials in their epidemiological context. Lancet. 1990 Apr 7;335(8693):827-38. doi: 10.1016/0140-6736(90)90944-z. PMID 1969567
- [Background] Wolf-Maier K, Cooper RS, Banegas JR, Giampaoli S, Hense HW, Joffres M, Kastarinen M, Poulter N, Primatesta P, Rodriguez-Artalejo F, Stegmayr B, Thamm M, Tuomilehto J, Vanuzzo D, Vescio F. Hypertension prevalence and blood pressure levels in 6 European countries, Canada, and the United States. JAMA. 2003 May 14;289(18):2363-9. doi: 10.1001/jama.289.18.2363. PMID 12746359
- [Background] Kearney PM, Whelton M, Reynolds K, Muntner P, Whelton PK, He J. Global burden of hypertension: analysis of worldwide data. Lancet. 2005 Jan 15-21;365(9455):217-23. doi: 10.1016/S0140-6736(05)17741-1. PMID 15652604
- [Background] Bray EP, Holder R, Mant J, McManus RJ. Does self-monitoring reduce blood pressure? Meta-analysis with meta-regression of randomized controlled trials. Ann Med. 2010 Jul;42(5):371-86. doi: 10.3109/07853890.2010.489567. PMID 20504241
- [Background] Fahey T, Schroeder K, Ebrahim S. Interventions used to improve control of blood pressure in patients with hypertension. Cochrane Database Syst Rev. 2005 Jan 25;(1):CD005182. doi: 10.1002/14651858.CD005182. PMID 15654709
- [Background] Ogedegbe G, Schoenthaler A. A systematic review of the effects of home blood pressure monitoring on medication adherence. J Clin Hypertens (Greenwich). 2006 Mar;8(3):174-80. doi: 10.1111/j.1524-6175.2006.04872.x. PMID 16522994
- [Background] AbuDagga A, Resnick HE, Alwan M. Impact of blood pressure telemonitoring on hypertension outcomes: a literature review. Telemed J E Health. 2010 Sep;16(7):830-8. doi: 10.1089/tmj.2010.0015. PMID 20815751
- [Derived] Bilger M, Koong AYL, Phoon IKY, Tan NC, Bahadin J, Bairavi J, Batcagan-Abueg APM, Finkelstein EA. Wireless Home Blood Pressure Monitoring System With Automatic Outcome-Based Feedback and Financial Incentives to Improve Blood Pressure in People With Hypertension: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Jun 9;10(6):e27496. doi: 10.2196/27496. PMID 34106085